CLINICAL TRIAL: NCT02865421
Title: Adipose Tissue Derived Stem Cell Based Hair Restoration Therapy for Androgenetic Alopecia
Acronym: AGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Mahmood S Choudhery, Assistant Professor, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: King Edward Medical University
Record Dates: First submitted 2016-06-21; First posted 2016-08-12 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Combination of SVF and PRP for Androgenetic Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stem cells (Experimental): adipose tissue derived stromal vascular fraction was used
  Interventions: Drug: stem cells
- platelet rich plasma (Experimental): platelet rich plasma isolated after centrifugation from the pt was transplanted
  Interventions: Drug: platelet rich plasma

INTERVENTIONS:
Drug: stem cells — adipose tissue derived stromal vascular fraction
  Other Names: stromal vascular fraction
  Arms: Stem cells
Drug: platelet rich plasma — platelet rich plasma transplanted in bald area at a distance
  Arms: platelet rich plasma

SUMMARY:
Androgenetic alopecia (AGA) is a common form of hair loss in both men and women, characterized by progressive patterned loss of hair from the scalp. The current study has been designed for restoration of hair in AGA by using a combination of stromal vascular fraction (derived from the adipose tissue) and human platelet rich plasma.

DETAILED DESCRIPTION:
Androgenetic alopecia (AGA) is a common form of hair loss in both men and women, characterized by progressive patterned loss of hair from the scalp. The prevalence of AGA increases significantly with age, 30% to 50% men are affected by the age of 30 and 50 years, respectively. 3 Further, women also suffer from different degrees of alopecia, 50% women are affected by the age of 60. AGA becomes a medical problem when the hair loss is subjectively considered as excessive, premature and distressing. Current treatment options for AGA include medications such as finasteride, dutasteride, spironolactone, flutamide, minoxidil etc. However, these medicines are suitable either for men or women only or they can only maintain existing hair but have no effect on hair regeneration. In addition treatment is expensive and requires prolonged usage of drugs, and if treatment is stopped any benefits gained will be lost. Therefore, a better solution is required that can stimulate the hair follicles to promote hair restoration in both sexes with long lasting effects. Recently, stem cell based therapies have revolutionized the field of regenerative medicine by providing treatment options for several diseases and disorders.

The current study has been designed for restoration of hair in AGA by implanting a combination of stromal vascular fraction (derived from the adipose tissue) and human platelet rich plasma.

The growth of human hair is an extremely complex process. Hair growth begins under the skin in structures called hair follicles. In AGA the size of hair follicles decreases due to loss of hair follicle stem or progenitor cells as a result hair follicles become inactive. Due to the inactivation of hair follicles large, pigmented terminal hairs are replaced by barely visible and de-pigmented vellus hairs. External factors can stimulate inactive hair follicles, as a result hair growth cycle can begin. other studies indicate that proteins and growth factors released by stem cells can play an important role in hair growth cycle. Considering these facts, current study has been designed as a possibility in the treatment of AGA by using a combination of autologous SVF and platelet rich plasma. In the current study,SVF derived from adipose tissue will be applied to restore hair growth.

Further, stem cells may also secrete various growth factors which can perform several functions including hair follicle stimulation.

Conventional approaches for hair refurbishment include medication and hair follicle transplantation surgery. However, these strategies are mostly ineffective in patients due to drawbacks including high cost, several side effects, unsatisfactory results, requirement for long lasting use of medicines and their efficacy is limited to either males or females. Therefore, contemporary therapies with promising results are required that should be effective in both sexes and outcomes should be long lasting. Stromal vascular fraction(SVF) based treatment for AGA can open a new avenue for the development of therapies for hair restoration. SVF can have multiple effects on miniaturized hair follicles by homing to the hair follicles and by their paracrine effects. The study will not only help the patients with hair loss but will also promote stem cell based regenerative medicine research in Pakistan by providing promising results.

ELIGIBILITY:
Inclusion Criteria:

* Patients 15 year or older
* Both males and females
* Patients diagnosed as male AGA, type III to VI using Hamilton - Norwood classification, as female pattern hair loss type I-III using Ludwig classification
* Active hair loss within last 12 months.
* Patients receiving fitness certificate from fitness committee (Medical Specialist, Plastic Surgeon and Anesthetist)

Exclusion Criteria:

* Pregnancy
* Diabetes
* Malignancy
* Global scalp hair thinning including occipital areas
* Patients with scalp inflammation, scalp infection (bacterial, viral, fungal and protozoal)
* Patients on anticoagulant therapy
* Patient on chemotherapy during the last five years

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
pull test | 6 months
  Approximately 20-60 hairs were grasped between the thumb, index and middle fingers from the base of the hairs near the scalp and firmly, but not forcefully, tugged away from the scalp.

SECONDARY OUTCOMES:
Trichoscan | 6 months
  Trichoscan is a method which combines standard epiluminescence microscopy with automatic digital image analysis for the measurement of all important hair parameters in situ.

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reid EE, Haley AC, Borovicka JH, Rademaker A, West DP, Colavincenzo M, Wickless H. Clinical severity does not reliably predict quality of life in women with alopecia areata, telogen effluvium, or androgenic alopecia. J Am Acad Dermatol. 2012 Mar;66(3):e97-102. doi: 10.1016/j.jaad.2010.11.042. Epub 2011 May 24. PMID 21601948